CLINICAL TRIAL: NCT06250855
Title: At Least One-year Long-term Clinical Outcomes Following Monofocal Toric Intraocular Lens Implantation: Observational Prospective Clinical Investigation
Brief Title: Observational Prospective Clinical Investigation on Monofocal Toric Intraocular Lens
Status: Completed | Type: Observational
Sponsor: SIFI SpA (Industry)
Responsible Party: Sponsor
Other Study IDs: 055/SI
Record Dates: First submitted 2024-02-01; First posted 2024-02-09 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Cataract; Astigmatism
Keywords: Cataract; Astigmatism; Monofocal IOL; Toric IOL
MeSH Terms: conditions — Cataract; Astigmatism

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Mini Toric IOL — Adults (males and females) ≥18 years with cataract and pre-existing corneal astigmatism who have undergone monocular or binocular Mini Toric Ready implantation after cataract surgery in which the cataract lens was removed by phacoemulsification, with circular capsulorhexis, leaving the posterior capsule intact.

SUMMARY:
Evaluation, at least one-year long-term, of the clinical performance and safety of Mini Toric Ready Intraocular Lens (IOL), a monofocal toric intraocular lens.

DETAILED DESCRIPTION:
Observational prospective clinical investigation based on the medical records of patients who undergone uncomplicated cataract surgery with implantation of Mini Toric Ready IOL and on a clinical visit after at least one year from the surgery. Eyes with corneal astigmatism ≥0.75 diopters were included. Postoperative evaluations included monocular or binocular uncorrected and corrected distance visual acuity; contrast sensitivity measured after at least one-year postoperatively.

ELIGIBILITY:
Inclusion Criteria:

* Eighteen years of age or older at the time of surgery and diagnosed with unilateral or bilateral cataracts;
* Preoperative total corneal astigmatism ≥0.75D;
* Unilateral or bilateral cataract removal by phacoemulsification;
* Clear intraocular media other than cataract;
* Willing and able to complete all required postoperative visits;
* Able to comprehend and sign a statement of informed consent consistent with local regulation for research in human subjects.

Exclusion Criteria:

* Subjects participating in a concurrent clinical trial or if they have participated in an ophthalmology clinical trial within the last 30 days before the surgery.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults (males and females) ≥18 years with cataract and pre-existing corneal astigmatism who have undergone monocular or binocular Mini Toric Ready implantation. Subjects enrolled in the investigation underwent cataract surgery in which the cataract lens was removed by phacoemulsification, with circular capsulorhexis, leaving the posterior capsule intact.
Sampling Method: Non-Probability Sample
Enrollment: 105 (Actual)
Dates: Start 2024-04-24 (Actual); Primary Completion 2024-10-27 (Actual); Study Completion 2024-10-27 (Actual)

PRIMARY OUTCOMES:
Evaluation of the Visual Performance | From 12 to 24 months post-surgery
  Evaluate Mini Toric Ready Intraocular Lens (IOL) performance in terms of correction of spherical and cylindrical visual defects, corrected and uncorrected monocular and/or binocular distance visual acuity at least 12 months post implant.

SECONDARY OUTCOMES:
Evaluation of the Stability | From 12 to 24 months post-surgery
  Intraocular Lens (IOL) Rotation Stability

OTHER OUTCOMES:
Evaluation of the safety profile: Adverse Events (AEs) | From 12 to 24 months post-surgery
  Incidence of Adverse events such as Posterior Capsular Opacification (PCO)
Evaluation of the safety profile | From 12 to 24 months post-surgery
  Rate of secondary surgical interventions (SSIs) related to the optical properties of the IOL after at least 12 months post implant.

CONTACTS AND LOCATIONS:
Locations (2):
- Romania (2):
  - Gauss Clinic Bacau, Bacau
  - Immunoeye SRL, Sfântu Gheorghe

IPD SHARING:
Plan to Share IPD: No